CLINICAL TRIAL: NCT02887989
Title: Immersive Virtual Reality Intervention for Non-Opioid Pain Management: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Brennan Spiegel, Director, Health Services Research, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045641
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Pain; Pain Management
Keywords: Virtual Reality; Non-Opioid Pain Management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality (Experimental): Patients will be allowed to use commercially-available VR equipment in their hospital rooms for up to 20 days, as needed to manage pain as an adjunct to opioid and non-opioid pain medication.
  Interventions: Device: Virtual Reality
- 'Health and Wellness Channel' (Sham Comparator): Patients will be allowed to watch relaxing television content in their hospital rooms for up to 20 days, as needed to manage pain as an adjunct to opioid and non-opioid pain medication.
  Interventions: Device: Health and Wellness Channel

INTERVENTIONS:
Device: Virtual Reality — A menu of VR experiences, lasting from 3-30 minutes each. For example, patients may watch a soothing virtual campfire, or fly over a scenic landscape, or play an interactive game.
  Arms: Virtual Reality
Device: Health and Wellness Channel — Relaxing content broadcast passively on the patient in-room television channel.
  Arms: 'Health and Wellness Channel'

SUMMARY:
The study is a randomized controlled trial (RCT) of VR non-opioid management vs. a control "sham" intervention for a broad and representative group of medical and surgical patients with pain. Hospitalized patients will receive specialized VR interventions, administered via portable VR headsets, to manage breakthrough pain. Control patients will view content on the in-room Health and Wellness television channel. Investigators will follow patients throughout the course of their hospitalization and monitor outcomes during and after their stays, including pain levels, medication requests, and quality of life.

DETAILED DESCRIPTION:
The study population will consist of 120 patients - 60 patients who are exposed to VR, and 60 control patients exposed to an audiovisual "sham" intervention. Investigators will select up to 120 hospitalized patients at CSMC admitted during the study period of November 2016 to September 2017. The inpatient wards serve patients ranging in age from 18 to over 100, allowing us to assess the feasibility of using VR across diverse age groups. Appropriate inpatients will be selected at random by Dr. Rosen or other authorized co-investigators or study staff, who will obtain relevant clinical variables from the EHR. All patients admitted to the hospital will be considered for the study. The location and identity of the inpatient will be relayed by their attending physician to a member of the study team, who will deliver a randomly selected intervention (either VR or Health and Wellness Channel) to the patient the same day (at the patient's discretion). The patient will continue usage as needed for up to 20 days of the hospital stay. VR Interventions include both relaxing environment and engaging games. The Health and Wellness Channel includes some of the same types of content, but it is delivered passively through the in-room television system. Investigators will examine changes in pain level, length of stay, medication requests (amount and timing), Quality of Life, Functioning, and Patient Satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the goals of the study and provide informed consent
* Any hospitalized patient under care of CSMC inpatient service (ISP), gastroenterology, or psychiatry, admitted between November 2016 and 30 September 2017, who is not excluded due to criteria listed below.
* At least one pain score ≥ 3 documented in the EHR.
* Received at least three doses of opioid medication for breakthrough pain, documented in the EHR.
* At least 18 years of age
* English speaking

Exclusion Criteria:

* Unable to consent to study due to cognitive difficulty
* Contact Isolation
* Current diagnosis of epilepsy, dementia, or other neurological disease that may prevent use of VR hardware and software
* Sensitivity to flashing light or motion
* Pregnancy, or a medical condition where the patient is prone to frequent nausea or dizziness
* Recent stroke
* Post-transplant patient, or pre-transplant patient with severe illness
* Patient on ventilator, BiPAP, or other breathing assistance equipment
* Injury to the eyes, face, neck, or arms that prevents comfortable use of VR hardware or software, or safe use of the hardware (e.g., open sores, wounds, or skin rash on face)
* Non-English speaking

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Spiegel, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654

RESULTS

PARTICIPANT FLOW:
Groups:
- In-Room Television: Patients will be allowed to watch relaxing television content in their hospital rooms for up to 20 days, as needed to manage pain as an adjunct to opioid and non-opioid pain medication.
  Health and Wellness Channel: Relaxing content broadcast passively on the patient in-room television channel.
Period: Overall Study
Arm/Group | Virtual Reality | In-Room Television
Started | 70 | 70
Completed | 61 | 59
Not Completed | 9 | 11
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality | In-Room Television | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Categorical [Count of Participants; unit: Participants] — Population: Rows differ due to uneven withdrawal and death.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 48 | 45 | 93
    >=65 years | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Rows differ due to uneven withdrawal and death
  years | 51.00 (15.09) | 50.02 (15.92) | 50.8 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Rows differ due to uneven withdrawal and death.
  Participants
    Female | 31 | 29 | 60
    Male | 30 | 30 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Rows differ due to uneven withdrawal and death
  Participants
    Race: white | 38 | 39 | 77
    Race: African-American | 21 | 10 | 31
    Race: Other | 2 | 10 | 12
Region of Enrollment [Number; unit: participants] — Rows differ due to uneven withdrawal and death
  participants
    United States | 61 | 59 | 120
Pain Type [Count of Participants; unit: Participants] — Population: Rows differ due to uneven withdrawal and death
  Participants
    Visceral | 23 | 20 | 43
    Somatic | 38 | 39 | 77
Last pain score pre-intervention [Mean (Standard Deviation); unit: units on a scale] — The primary outcome was pain intensity collected via ecological momentary assessment in the course of usual care by hospital staff. At three-to-four hour intervals during waking hours, subjects were asked by their assigned nurse to rate their pain using a standard 11-point numeric rating scale (NRS), where 0 is "no pain" and 10 is "worst imaginable pain." Population: Rows differ due to uneven withdrawal and death
  units on a scale | 3.31 (2.83) | 3.97 (3.13) | 3.63 (2.99)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Ratings (NRS)
Description: The primary outcome was pain intensity collected via ecological momentary assessment in the course of usual care by hospital staff. At three-to-four hour intervals during waking hours, subjects were asked by their assigned nurse to rate their pain using a standard 11-point numeric rating scale (NRS), where 0 is "no pain" and 10 is "worst imaginable pain." Data are summarized as pre/post mean and in time-series.
Time Frame: Approximately every 3-4 hours for the period 48 hours pre and post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality | In-Room Television
Number analyzed (Participants) | 61 | 59
score on a scale | 4.66 (2.91) | 4.94 (3.04)

2. Primary Outcome: Morphine Milligram Equivalents (MME)
Description: Opioid usage was defined as mean total milligrams of morphine equivalent (MME), calculated by first multiplying the quantity of each prescribed medication by the strength of that medication (milligrams of given opioid per unit dispensed), and then multiplying this quantity-strength product by conversion factors derived from published sources to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription. The mean pre-intervention MME for subjects in each arm was calculated by adding the morphine equivalents for each prescription dispensed during the 48 hours before intervention, while the post-intervention MME for subjects in each arm was calculated by adding the morphine equivalents for each prescription dispensed during the 48 hours after intervention.
Time Frame: assessed at 48 hours before intervention and 48 hours after intervention
Population: Not all patients received opioids
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents (MME)
Arm/Group | Virtual Reality | In-Room Television
Number analyzed (Participants) | 48 | 53
Morphine milligram equivalents (MME)
  pre-intervention MME | 75.07 (7.25) | 80.83 (6.86)
  post-intervention MME | 77.08 (6.34) | 81.04 (6.193888)
Statistical Analysis 1: Comparison: Virtual Reality vs In-Room Television; Test type: Superiority; p = .6570, t-test, 2 sided

3. Secondary Outcome: Length of Stay) LOS
Description: defined as the number of days from the date of admission to date of hospital discharge. Hour of admission was not available in these data, so patients admitted late on Day 0 (i.e., before midnight), and discharged the following calendar day (i.e., between 00:00 and 23:59), were counted as a 1-day hospital stay. Patients who were admitted and discharged on the same calendar day were considered to have an LOS of 0.
Time Frame: Count of Days in Hospital Stay up to 20
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Virtual Reality | In-Room Television
Number analyzed (Participants) | 61 | 59
days | 5.11 (.58) | 5.64 (.95)
Statistical Analysis 1: Comparison: Virtual Reality vs In-Room Television; Test type: Superiority; p = .6339, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 96 hours
Arm/Group | Virtual Reality | In-Room Television
All-Cause Mortality (participants affected / at risk) | 1/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

LIMITATIONS AND CAVEATS:
Usage data was not collected, so no conclusions regarding actual dose/response can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02887989/Prot_SAP_000.pdf